CLINICAL TRIAL: NCT02693639
Title: Prediction Value of PANX1 in Infection Post Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lin Zhong (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor-Investigator, Lin Zhong, Director of department of liver transplantation, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: SHLTQC-1
Record Dates: First submitted 2016-02-17; First posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Infection
Keywords: PANX1; Infection; Liver transplantation
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- liver transplantation grafts

SUMMARY:
The purpose of this study is to determine prediction value of PANX1 expression in infection post liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent liver transplantation.

Exclusion Criteria:

* re-transplantation
* multiorgan transplantation
* living donors or split-liver donors liver transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent liver transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-02; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Post-transplant infections | 90 days
  Frequency of clinically or microbiologically documented infection after transplantation.